CLINICAL TRIAL: NCT04217954
Title: Hepatic Arterial Infusion Chemotherapy With Oxaliplatin, 5-fluorouracil and Bevacizumab Plus Intravenous Toripalimab for Advanced Biliary Tract Cancer
Brief Title: HAIC With Oxaliplatin, 5-FU and Bevacizumab Plus Intravenous Toripalimab for Advanced BTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Wang, MD, Professor, Peking University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FIBTC
Record Dates: First submitted 2020-01-01; First posted 2020-01-06 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: hepatic arterial infusion chemotherapy; oxaliplatin; 5-fluorouracil; bevacizumab; Toripalimab; advanced biliary tract cancer
MeSH Terms: interventions — Fluorouracil; Bevacizumab; toripalimab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OXA, 5-FU and Bev plus Toripalimab (Experimental): the patients enrolled in this arm would receive hepatic arterial infusion chemotherapy with oxaliplatin, 5-fluorouracil and bevacizumab plus intravenous Toripalimab
  Interventions: Drug: OXA, 5-FU and bevacizumab plus Toripalimab

INTERVENTIONS:
Drug: OXA, 5-FU and bevacizumab plus Toripalimab — 1. concomitant treatment: A. HAIC: oxaliplatin (40 mg/m2 for 2 hours), 5-fluorouracil (800 mg/ m2 for 22 hours) on days 1-3, and arterial bevacizumab 300mg for 2 hours on d1 before oxaliplatin through a percutaneously implanted port-catheter system.
     B. Intravenous PD-1 inhibitor (Toripalimab) 240 mg for 30-60 minutes on d1 before the HAIC.
     The concomitant treatment repeat every three week, up to 6 cycles.
  2. Maintenance treatment: Bevacizumab (300mg) + PD-1 inhibitor (Toripalimab 240mg) will be given intravenously, every 3 weeks.
  Other Names: FOLFOX

SUMMARY:
Hepatic arterial infusion chemotherapy (HAIC) deliver high concentration of chemotherapeutic agents directly to the liver tumor, was proved to be effective for intrahepatic and perihilar cholangiocarcinoma. Based on the potential synergistic effect of bevacizumab, chemotherapy and PD-1 inhibitor, this phase II clinical study want to test the efficacy and safety using intra-arterial infusion of oxaliplatin, 5-fluorouracil and bevacizumab combined with intravenous infusion of PD-1 inhibitor (Toripalimab) in the treatment of unresectable biliary malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Biliary tract cancer proved by histology or cytology
2. Metastatic advanced or locally advanced unresectable biliary tract cancer, including gallbladder cancer, intrahepatic cholangiocarcinoma and perihilar cholangiocarcinoma, decided by hepatobiliary doctor and radiologist.
3. At least one measurable lesion within liver;
4. No prior intra-arterial/systemic chemotherapy or other systemic therapies
5. Prior resection, TACE or ablation will be allowed.
6. Age from 18 years old to 80 years old.
7. the performance of Eastern Cooperative Oncology Group (ECOG) <2
8. Child-Pugh A or Child-Pugh B (≤ score 7).
9. Expectant survival time ≥ 3 months.
10. Baseline blood count test and blood biochemical must meet following criteria:

    1. Hemoglobin ≥ 90 g/L;
    2. Absolute neutrophil count ≥ 1.5×10^9/L;
    3. Blood platelet count ≥ 100×10^9/L;
    4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times of upper limit of normal (ULN);
    5. Total bilirubin ≤ 2 times of ULN;
    6. Serum creatinine ≤ 1.5 times of ULN;
    7. Albumin ≥ 30 g/L.
11. Patients sign informed consent.

Exclusion Criteria:

1. Distal cholangiocarcinoma.
2. Allergic to contrast agent.
3. Pregnant or lactational.
4. Allergic to 5-fluorouracil, or have metabolic disorder of 5-fluorouracil.
5. More than 80 years old.
6. Previous systematic chemotherapy or radiotherapy.
7. Child-Pugh C or Child-Pugh B (≥ score 8).
8. Coinstantaneous a lot of malignant hydrothorax or ascites.
9. History of organ transplantation (including bone marrow auto-transplantation and peripheral stem cell transplantation).
10. Coinstantaneous infection and need anti-infection therapy.
11. Hepatitis B virus DNA load ≥ 100 IU/ml (patients whose hepatitis B virus DNA load decreased to < 100 IU/ml after anti-virus therapy could be enrolled).
12. Coinstantaneous peripheral nervous system disorder or with history of obvious mental disorder and central nervous system disorder.
13. Diagnosed other kinds of malignant within 5 years, except for non-melanoma skin cancer and carcinoma in situ of cervix.
14. Without legal capacity.
15. Impact the study because of medical or ethical reasons.
16. Uncorrectable coagulation disorder.
17. Obvious abnormal in ECG or obvious clinical symptoms of heart disease, like congestive heart failure (CHF), coronary heart disease with obvious clinical symptoms, unmanageable arrhythmia and hypertension.
18. History of myocardial infarction within 12 months, or Grade III/IV of heart function.
19. Severe liver disease (like cirrhosis), renal disease, respiratory disease, unmanageable diabetes or other kinds of systematic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | From the start of treatment until the end of treatment, up to approximately 3 years
  CR plus PR according to imRECIST

SECONDARY OUTCOMES:
Overall survival | From the start of treatment until death or lost to follow-up, up to approximately 3 years
  date from the start of treatment until death or lost to follow-up, whichever happen first, assessed at least 6 months
Adverse events | From the start of treatment until the end of treatment, up to approximately 3 years
  type and incidence of adverse events
Progression-free survival | From the start of the treatment until first documented progression or death from any cause, whichever came first, assessed up to approximately 3 yearsse date of disease progression
  date from the first treatment to the date of disease progression, lost to follow-up or death, whichever happen first

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, MD, Study Director — Department of Interventional Therapy, Peking University Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
signed informed consent with patients

REFERENCES:
- [Background] Park J, Kim MH, Kim KP, Park DH, Moon SH, Song TJ, Eum J, Lee SS, Seo DW, Lee SK. Natural History and Prognostic Factors of Advanced Cholangiocarcinoma without Surgery, Chemotherapy, or Radiotherapy: A Large-Scale Observational Study. Gut Liver. 2009 Dec;3(4):298-305. doi: 10.5009/gnl.2009.3.4.298. Epub 2009 Dec 31. PMID 20431764
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Boehm LM, Jayakrishnan TT, Miura JT, Zacharias AJ, Johnston FM, Turaga KK, Gamblin TC. Comparative effectiveness of hepatic artery based therapies for unresectable intrahepatic cholangiocarcinoma. J Surg Oncol. 2015 Feb;111(2):213-20. doi: 10.1002/jso.23781. Epub 2014 Sep 1. PMID 25176325
- [Background] Wang X, Hu J, Cao G, Zhu X, Cui Y, Ji X, Li X, Yang R, Chen H, Xu H, Liu P, Li J, Li J, Hao C, Xing B, Shen L. Phase II Study of Hepatic Arterial Infusion Chemotherapy with Oxaliplatin and 5-Fluorouracil for Advanced Perihilar Cholangiocarcinoma. Radiology. 2017 May;283(2):580-589. doi: 10.1148/radiol.2016160572. Epub 2016 Nov 7. PMID 27820684
- [Background] Gao F, Yang C. Anti-VEGF/VEGFR2 Monoclonal Antibodies and their Combinations with PD-1/PD-L1 Inhibitors in Clinic. Curr Cancer Drug Targets. 2020;20(1):3-18. doi: 10.2174/1568009619666191114110359. PMID 31729943
- [Background] Hegde PS, Wallin JJ, Mancao C. Predictive markers of anti-VEGF and emerging role of angiogenesis inhibitors as immunotherapeutics. Semin Cancer Biol. 2018 Oct;52(Pt 2):117-124. doi: 10.1016/j.semcancer.2017.12.002. Epub 2017 Dec 8. PMID 29229461
- [Background] Mathew M, Enzler T, Shu CA, Rizvi NA. Combining chemotherapy with PD-1 blockade in NSCLC. Pharmacol Ther. 2018 Jun;186:130-137. doi: 10.1016/j.pharmthera.2018.01.003. Epub 2018 Jan 31. PMID 29352857
- [Background] Dalgleish AG. Rationale for combining immunotherapy with chemotherapy. Immunotherapy. 2015;7(3):309-16. doi: 10.2217/imt.14.111. PMID 25804482
- [Background] Longo V, Brunetti O, Azzariti A, Galetta D, Nardulli P, Leonetti F, Silvestris N. Strategies to Improve Cancer Immune Checkpoint Inhibitors Efficacy, Other Than Abscopal Effect: A Systematic Review. Cancers (Basel). 2019 Apr 15;11(4):539. doi: 10.3390/cancers11040539. PMID 30991686